CLINICAL TRIAL: NCT06139393
Title: Study on Efficacy and Safety of HR091506 Tablets in Treatment of Gout With Hyperuricemia in Adults
Brief Title: Clinical Study of HR091506 Tablets in Treatment of Gout With Hyperuricemia in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR091506-302
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Gout With Hyperuricemia in Adults
MeSH Terms: interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A: HR091506 tablets + placebo of febuxostat tablets (Experimental)
  Interventions: Drug: HR091506 tablets + placebo of febuxostat tablets
- Treatment group B: febuxostat tablets + placebo of HR091506 tablets (Active Comparator)
  Interventions: Drug: febuxostat tablets + placebo of HR091506 tablets

INTERVENTIONS:
Drug: HR091506 tablets + placebo of febuxostat tablets — HR091506 tablets 20mg qd + placebo of febuxostat tablets 20mg qd from Week 1 to 4, HR091506 tablets 40mg qd + placebo of febuxostat tablets 40mg qd from Week 5 to 28.
  Arms: Treatment group A: HR091506 tablets + placebo of febuxostat tablets
Drug: febuxostat tablets + placebo of HR091506 tablets — febuxostat tablets 20mg qd + placebo of HR091506 tablets 20mg qd from Week 1 to 4, febuxostat tablets 40mg qd + placebo of HR091506 tablets 40mg qd from Week 5 to 28.
  Arms: Treatment group B: febuxostat tablets + placebo of HR091506 tablets

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of HR091506 tablets for treatment of gout with hyperuricemia in adults, and to compare the results with febuxostat tablets in the same doses.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, male or female;
2. BMI: 18.0-30.0 kg/m2;
3. Meet the 2015 ACR/EULAR gout classification criteria;
4. Fast serum uric acid ≥ 480 μmol/L on 2 different days during the screening perid;
5. Willing to ues contraceptive measures during the study;
6. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. History of acute gout attack within 4 weeks before randomization.
2. Subjects who have undergone major surgery or organ transplantation within 3 months before randomization.
3. Subjects with major cardiovascular disease within 6 months before randomization.
4. History of chronic infection or recurrent infection within 1year before randomization.
5. History of malignant tumor or current history of combined malignant tumor within 5 years before screening.
6. History of secondary hyperuricemia, refractory gout, or xanthine metabolism disorder.
7. Subjects with poorly controlled blood pressure or diabetes mellitus.
8. History of chronic diffuse connective tissue disease and/or massively elevated urate diseases and/or untreated clinically significant thyroid disease.
9. History of diseases that may affect the in vivo process, safety evaluation, or subjects' participation in the research.
10. Abnormal laboratory tests that may affect subjects participating in the research.
11. Combined use of prohibited drugs.
12. Allergic to ingredient or component of the experimental drug.
13. Participated in other clinical trials within 1 month before randomization.
14. Pregnant or nursing women.
15. History of drug abuse, drug use and/or excessive drinking within 1 year before screening.
16. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with serum uric acid level < 360 μmoL/L at Week 28 | Week 28

SECONDARY OUTCOMES:
Proportion of subjects with serum uric acid level < 360 μmol/L at each visit. | at week 4,8,12,16,20and24 after administration
Proportion of subjects with serum uric acid level < 300 μmol/L at each visit | at week 4,8,12,16,20,24and28 after administration
Change of serum uric acid level from baseline to every visit | at week 4,8,12,16,20,24 and28 after administration
Proportion of subjects with ≥1 gout flare during treatment stage | during treatment stage

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided